CLINICAL TRIAL: NCT04178889
Title: Second Primary Lung Cancer Cohort Study (SPORT)
Acronym: SPORT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Cancer Research UK (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: P02514
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be processed and separated into various components for storage, before batched analysis.
  Consent will be sought for the sample components to be kept for up to 15 years following the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who have had curative treatment for lung cancer are at an increased risk of developing second primary lung cancers (and other cancers) over the next 10 years. Doctors need to develop better ways of monitoring patients during follow up so we can intervene as quickly as possible with further treatments. Measuring DNA in the blood which has come from the tumour, so called circulating tumour DNA (ctDNA), may be one way to do this.

DETAILED DESCRIPTION:
This is a multi-centre, observational basic science study to follow patient who have undergone radical treatment, surgery or radiotherapy for Non-small Cell Lung Cancer (NSCLC) between two and five years previously. Following consent, participants will be asked to provide blood samples every six months for up to the next five years. Information from their routine clinical care, including information from any imaging, diagnostic tissue samples and blood tests will be collected. We will also request access to any original surplus diagnostic material, as well as future, excess tissue from diagnostic samples.

Blood samples will be analysed using various new scientific techniques looking to correlate emergence of new primary cancer (or recurrence of original NSCLC) with blood based markers.

ELIGIBILITY:
Inclusion Criteria:

* previous treatment with curative intent (surgery or radical (chemo)radiotherapy) for stage I-IIIA primary NSCLC
* at least two years post first treatment date of first primary NSCLC
* able to provide informed consent

Exclusion Criteria:

* Primary lung tumour was a carcinoid tumour
* in the opinion of the managing clinician, thought unlikely to survive 12 months from time of potential recruitment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been treated with curative intent (surgery/(chemo)radiotherapy) for stage I to IIIA Non-small cell carcinoma, between two and five years ago.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment of 850 patients who have undergone treatment with curative intent for stage 1 - 3A non-small cell lung cancer. | 5 years
  In order to:
  collect baseline demographics, clinical and past medical history to obtain blood samples every 6 months after recruitment
  to collect relevant imaging and clinical data as part of their on-going routine clinical care

SECONDARY OUTCOMES:
To collect blood samples from the cohort of patients. | From recruitment through to end of study (or 5 year follow up point, whichever comes first)
  Have the blood samples been collected at follow up visits.
To collect surplus diagnostic tissue from the cohort of patients. | Identify original diagnostic sample at recruitment.
  To collect surplus diagnostic tissue from original non-small cell lung cancer.
To collect surplus diagnostic tissue from new cancer occurrences or relapse from the cohort of patients | From recruitment to end of study (or 5 year follow up point, whichever comes first)
  Collection of surplus diagnostic tissue if any second primary cancer or recurrence occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rintoul, PhD FRCP, Principal Investigator — Royal Papworth Hospital NHS Trust
Locations (1):
- Royal Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The only clinical data available to researchers will be anonymised. Permission will be sought at consent to retain data sets for up to 15 years at the end of the study to use for this study or other ethically approved studies.

REFERENCES:
- [Background] Barclay ME, Lyratzopoulos G, Walter FM, Jefferies S, Peake MD, Rintoul RC. Incidence of second and higher order smoking-related primary cancers following lung cancer: a population-based cohort study. Thorax. 2019 May;74(5):466-472. doi: 10.1136/thoraxjnl-2018-212456. Epub 2019 Feb 18. PMID 30777897
- [Background] Wan JCM, Massie C, Garcia-Corbacho J, Mouliere F, Brenton JD, Caldas C, Pacey S, Baird R, Rosenfeld N. Liquid biopsies come of age: towards implementation of circulating tumour DNA. Nat Rev Cancer. 2017 Apr;17(4):223-238. doi: 10.1038/nrc.2017.7. Epub 2017 Feb 24. PMID 28233803